CLINICAL TRIAL: NCT05800132
Title: Évaluation de la Performance Diagnostique du dépistage du Cancer du Sein, Pour Une Seconde Lecture Des clichés de Mammographie assistée du Dispositif médical à Base d'Intelligence Artificielle MammoScreen
Brief Title: Diagnostic Performance of Breast Cancer Screening Second Reading Process Assisted by AI
Acronym: IMA-L2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Therapixel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: ID-RCB 2022-A01488-35
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: artificial intelligence; breast cancer screening; second reading
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L2 - Standard second read (No Intervention): Interpretation of mammograms done by a radiologist accredited to do second reading in France.
- L2-AI - AI-assisted second read (Experimental): Interpretation of mammograms done by the AI-based device. Mammograms deemed suspicious by the AI (i.e., receiving an AI global score higher than a defined threshold) will be interpreted by a radiologist accredited to do second reading in France. Mammograms assessed as negative or low suspicious by the AI won't be further interpreted by a radiologist.
  Interventions: Device: MammoScreen

INTERVENTIONS:
Device: MammoScreen — Diagnostic reading aid for breast cancer screening
  Arms: L2-AI - AI-assisted second read

SUMMARY:
The goal of this clinical trial is to compare, for the second reading of screening mammograms, the standard of care with an AI assisted scenario.

The main questions it aims to answer are:

* will the experimental pathway be non-inferior to the standard pathway?
* will the experimental pathway be economically superior to the standard pathway?

Participants will receive screening mammograms, as part of the breast cancer screening program. Researchers will compare the interpretation made by the second reader in the standard pathway with the AI assisted interpretation made by a different reader in the experimental pathway.

DETAILED DESCRIPTION:
All mammograms eligible for a second reading, and included in the study, go through 2 arms:

* Conventional second reading by a radiologist accredited to do second reading in France (L2 control arm),
* Second reading assisted by the AI (L2-AI experimental arm): mammograms will be read by the AI first and only if deemed suspicious, a radiologist accredited to do second reading in France will review them.

The most pejorative assessment among the two arms is used as the final decision: if both arms consider the mammogram as negative, the participant won't be recalled, if one arm consider the mammogram as positive, the participant will be called back for further examinations.

Clinical performances and economical impacts of both scenarii will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to the French social security system
* Whose mammograms meet the following characteristics: 4 (2 per breast, CC and MLO) meeting local regulatory standards and with correct DICOM metadata,
* Whose mammograms have been determined to be normal or to have benign lesions by the radiologist who performed the first reading of the images (L1) in the framework of the organized breast cancer screening program
* Having expressed her willingness to participate in the study, to undergo all the procedures and to make herself available for the expected duration of their participation,
* Having completed and signed the informed consent form.

Exclusion Criteria:

* Woman with breast implants,
* With clinical symptoms of breast cancer,
* With a history of breast surgery (breast reduction or surgery for benign lesion),
* Pregnant or breastfeeding,
* With medical conditions that may interfere with her ability to understand the requirements of the protocol or give informed consent,
* Deprived of liberty by judicial or administrative order,
* Participant whose mammogram images have at least one of the following defects: poor quality of the images, non-standard mammography (projection, magnification, compression), ML/LM/SIO/XCCL or XCCM view.

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Recall rate | End of the inclusion period 24 months
  Number of patients that are called back for further examinations divided by the total number of patient receiving a second reading.

SECONDARY OUTCOMES:
Cancer detection rate | End of the inclusion period 24 months
  Number of biopsy proven cancers divided by the total number of patient receiving a second reading
Sensitivity and Specificity | End of the follow_up period 48 months
  True and false-positive rate
Economic impact | End of the follow_up period 48 months
  Difference in direct medical costs between the two arms Difference in annual budgetary impact on the French National Health Insurance between the two arms
Time-to-results | End of the inclusion period 24 months
  Time period [in days] between the day of the screening and the access to results
Reading time | End of the inclusion period 24 months
  Time needed [in seconds] to interpret a mammogram

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Seradour, Principal Investigator — Centre Régional de Coordination des Dépistages des Cancers (CRCDC) Région Sud PACA
Locations (7):
- France (7):
  - Centre de radiologie Les Défensions, Aubagne
  - Var Imagerie Medicale, Draguignan
  - VAR IMAGERIE MEDICALE - Centre d'Imagerie Médicale Le Clipper, Fréjus
  - VAR IMAGERIE MEDICALE - Clinique Les Lauriers, Fréjus
  - Cabinet de Radiologie du Cabot, Marseille
  - Centre de Sénologie Mermoz, Marseille
  - VAR IMAGERIE MEDICALE - Centre d'Imagerie Médicale Epsilon, Saint-Raphaël

IPD SHARING:
Plan to Share IPD: No